CLINICAL TRIAL: NCT02236286
Title: Frontal Cortex and Gait Freezing in Parkinson's Disease: Rehabilitation Impact
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Fay B. Horak, Professor of Neurology, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 8979
Record Dates: First submitted 2014-09-03; First posted 2014-09-10 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Parkinson's Disease
Keywords: freezing of gait (FOG); balance; gait; exercise
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): Subjects will participate in a 90-minute, group (6 per group) exercise session 3 days per week for 6 weeks (18 sessions). The theoretical basis for our novel Agility Boot Camp (ABC) exercise program is based on research that identified the primary neurophysiological and cognitive constraints that limits balance and mobility in PD. The exercises are designed as a circuit with several types of movement-skills specifically focused on improving different postural domains with cognitive challenges such as memorized sequences and dual tasking.
  Interventions: Behavioral: Exercise
- Chronic Disease Management Education (Active Comparator): Subjects will also receive (cross-over) six weeks of educational classes. The Education program will teach subjects, chronic disease self-management - how to live better with their parkinsonism. Classes will consist of 6 subjects per group meeting for 90 minute sessions, once a week for six weeks. Subject will do an additional 120 minutes of relaxation at home/week.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Agility Boot Camp (ABC) exercise intervention consisting of 18 sessions of group exercise led by an exercise trainer.

SUMMARY:
This project will relate our new quantification of Freezing of Gait (FoG) in Parkinson's disease, using body worn inertial sensors (Aim I), with abnormalities in state-of-the-art, resting state, functional brain connectivity (Aim II), and determine the number of subjects needed for a future, randomized clinical trial to test the efficacy of our novel, Agility Boot Camp (ABC) rehabilitation intervention for FoG (Aim III). The technological approaches to these aims are cutting edge and will allow us to develop sensitive behavioral and brain biomarkers for gait disorders in Parkinson's disease (PD) for use in future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50-90 years old.
* No musculoskeletal or peripheral or central nervous system disorders (other than idiopathic Parkinson disease, iPD) that could significantly affect balance or gait .
* Capable of following directions.
* iPD subjects: United Kingdom Brain Bank criteria, i.e., bradykinesia and at least one of the following: rest tremor, muscular rigidity, and postural instability not cause by visual, vestibular, cerebellar or proprioceptive dysfunction. Unilateral onset, response to levodopa.

Exclusion Criteria:

* Inability to stand or walk for 2 min without an assistive device
* Recent changes in medication
* Excessive use of alcohol or recreational drugs,
* Contraindications to MRI scans (eg, claustrophobia, metal in body)
* Intervention subjects will be excluded if: 1) participating in a vigorous exercise program more than 2 x/week, 2) A medical condition that contraindicates exercise participation.
* Idiopathic PD subjects: Same as above and deep brain stimulation electrodes. Significant tremor that would interfere with MRI scan.

Control subjects:

* Will be matched for age and gender to iPD group.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-09; Primary Completion 2018-09 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Change in Freezing of Gait Index | Three timepoints; baseline, 6 weeks (after Arm 1), 12 weeks (after Arm 2)
  Quantify amount of freezing in the legs ('trembling of knees'), defined as the square of the total power in the 3-8 Hz band, divided by the square of the total power in the 0.5-3 Hz band.

SECONDARY OUTCOMES:
Change in the New Freezing of Gait Questionnaire (NFOGQ) score | Three timepoints; baseline, 6 weeks (after Arm 1), 12 weeks (after Arm 2)
  The NFOGQ will be used to identify 'freezers' (score > 3). It is a self-report measure that begins with the presentation of a short video to illustrate FoG during walking, turning and starting gait and then follows with questions related to frequency and duration of each type of FoG episode.
Change in PDQ-39 score | Three timepoints; baseline, 6 weeks (after Arm 1), 12 weeks (after Arm 2)
  The Parkinson's Disease Quality of Life Questionnaire (PDQ-39) has 39 questions reflecting eight domains of quality of life (Mobility, Activities of Daily Living, Emotional well-being, Stigma, Social Support, Cognition, Communication, and Bodily Discomfort). Each item scores from 0 (never) to 4 (always). Subscale scores and a summary index representing the global health-related quality of life will be calculated, with higher scores representing worse quality of life. Convergent validity is very good and discriminative validity for PD severity levels have been established. The PDQ-39 will reflect limitations to participation in community mobility.
Change in Activities of Balance Confidence (ABC) Questionnaire score | Three timepoints; baseline, 6 weeks (after Arm 1), 12 weeks (after Arm 2)
  ABC questionnaire consists of 16 questions about how balance confidence limits participating in the community such as riding an escalator or walking in a crowded area, Subjects indicate their confidence from 0 - 100% in being able to complete each of the tasks. A score of 80% indicates an average level of physical functioning for older adults.
Change in instrumented gait and balance measures | Three timepoints; baseline, 6 weeks (after Arm 1), 12 weeks (after Arm 2)
  Gait: Walking metrics will be collected during short (7 meter, 180° turn, 7 meter) and long (2 minutes) walks.
  Instrumented Brief BESTest - another variation of the BESTest (Balance Evaluation - Systems Test) that will be administered with inertial sensors to quantify the important metrics of the test.
Change in mini-BESTest score | Three timepoints; baseline, 6 weeks (after Arm 1), 12 weeks (after Arm 2)
  The mini-BESTest assesses dynamic balance via a 14-item test that measure multiple domains of balance including anticipatory postural adjustments, reactive postural control, sensory orientation, and dynamic gait.
Change in UPDRS score | Three timepoints; baseline, 6 weeks (after Arm 1), 12 weeks (after Arm 2)
  The Unified Parkinson's Disease Rating Scale (UPDRS) Motor Subscale is a 10-minute assessment of motor signs related to severity of PD. If the investigators have trouble recruiting subjects of similar severity in the 2 groups (PD Freezers and Non-Freezers, then they will use the Postural Instability and Gait Disability (PIGD) Subscore as a covariate in data analysis.
Change in locomotor neural network functional connectivity strength | Three timepoints; baseline, 6 weeks (after Arm 1), 12 weeks (after Arm 2)
  Changes in resting state blood oxygen level dependent neural signal synchronization between Supplementary Motor Area and Mesencephalic locomotor region across 3 time points.
Change in SCOPA-COG score | Three timepoints; baseline, 6 weeks (after Arm 1), 12 weeks (after Arm 2)
  Scales for Outcomes in Parkinson's Disease-cognition (SCOPA-COG) is an instrument that was designed to assess the specific 'frontal-subcortical' cognitive deficits found in Parkinson's disease. The scale, consisting of 10 items, covers the following domains: memory and recall (verbal recall, digit span backward, and indicate cubes), attention (counting backward, months backward), executive function (fist-edge-palm, semantic fluency, and dice), visual-spatial functions (assembly pattern), and memory (delayed recall). The score ranges from 0-43 points with higher scores reflecting better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Fay B Horak, PhD, PT, Principal Investigator — VA Portland Health Care System (VAPORHCS)
Locations (1):
- VA Portland Health Care System (VAPORHCS), Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886